CLINICAL TRIAL: NCT02079415
Title: Study of Outcome of Infants of Diabetic Mothers in a Tertiary Hospital Set up
Brief Title: Infants of Diabetic Mothers: A Cohort Study
Status: Completed | Type: Observational
Sponsor: Security Forces Hospital (Other)
Responsible Party: Principal Investigator, OMER B ABDELBASIT, Consultant Neonatolgist, Security Forces Hospital
Other Study IDs: OJS2817
Record Dates: First submitted 2014-02-16; First posted 2014-03-05 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Pregnancy in Diabetes; Fetal Complications
Keywords: NICU
MeSH Terms: conditions — Pregnancy in Diabetics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Prevention of complications in infants of diabetic mothers — strict glycemic control in diabetic pregnancies
  Other Names: Congenital malformations

SUMMARY:
Saudi Arabia has been named by the International Diabetes Federation as among the top ten countries with highest prevalence of diabetes. Women are said to have overall prevalence twice that for men. With high birth rate in the country we decided to look at the impact of diabetic pregnancies on their off-springs

DETAILED DESCRIPTION:
Diabetics are followed regularly in diabetic outpatient clinics where dietary and medical management are offered. Diabetic pregnancies are managed by a team consisting of diabetologist, obstetrician, feto-maternal obstetrician and dietician.

Management of these pregnancies depends on whether these women have pre-gestational or gestational diabetes. Very few diabetic women have exposure to preconceptual advice. For this reason we opted to find out the outcome of infants of diabetic mothers compared to those mothers who are essentially normal with no associated medical or obstetric disorders. Equally we wanted to see if there are differences in the outcome of infants born to pre-gestational and gestational diabetic mothers.

ELIGIBILITY:
Inclusion Criteria:All infants born to diabetic mothers

* Infants born to mothers with normal pregnancies

Exclusion Criteria:

* Infants born to mothers with other medical disorders before or during pregnancy which may affect the newborn

Min Age: 1 Hour | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All Infants of diabetic mothers born at security Forces Hospital, Riyadh
Sampling Method: Non-Probability Sample
Enrollment: 601 (Actual)
Dates: Start 2011-01; Primary Completion 2012-01 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Congenital malformations | At time of first clinical examination
  Assess presence of congenital malformations in infants of diabetic mothers

SECONDARY OUTCOMES:
Length of hospital stay | Until discharge from hospital or death
  To assess the length of hospital stay for infants of diabetic mothers

OTHER OUTCOMES:
Preterm birth | Immediately at day 1
  To assess incidence of preterm birth in infants of diabetic mothers
Admission to neonatal intensive care unit | day 1
  To assess the need of infants of diabetic mothers for admission to neonatal intensive care

CONTACTS AND LOCATIONS:
Overall Officials: ABEER E LASHEEN, MBBS, Study Director — Security Forces Hospital
Locations (1):
- Security Forces Hospital, Riyadh, Central, Saudi Arabia

REFERENCES:
- [Background] Alqurashi KA, Aljabri KS, Bokhari SA. Prevalence of diabetes mellitus in a Saudi community. Ann Saudi Med. 2011 Jan-Feb;31(1):19-23. doi: 10.4103/0256-4947.75773. PMID 21245594
- [Background] Persson M, Norman M, Hanson U. Obstetric and perinatal outcomes in type 1 diabetic pregnancies: A large, population-based study. Diabetes Care. 2009 Nov;32(11):2005-9. doi: 10.2337/dc09-0656. Epub 2009 Aug 12. PMID 19675195
- [Result] Yang J, Cummings EA, O'connell C, Jangaard K. Fetal and neonatal outcomes of diabetic pregnancies. Obstet Gynecol. 2006 Sep;108(3 Pt 1):644-50. doi: 10.1097/01.AOG.0000231688.08263.47. PMID 16946226